CLINICAL TRIAL: NCT05652517
Title: Image Fusion of Integrating Fluoroscopy Into 3D Computed Tomography in Guidance of Vein of Marshall Ethanol Infusion During Persistent Atrial Fibrillation Ablation
Brief Title: Univu-guided Vein of Marshall Ethanol Infusion (Marshall-Merge)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jian Sun, Principal investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-22-009
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopy-guided VOMEI (Active Comparator): Vein of Marshall ethanol infusion guided by fluoroscopy alone
  Interventions: Procedure: Vein of Marshall ethanol infusion
- UNIVU-guided VOMEI (Experimental): Vein of Marshall ethanol infusion guided by CARTO UNIVU and fluoroscopy
  Interventions: Procedure: Vein of Marshall ethanol infusion

INTERVENTIONS:
Procedure: Vein of Marshall ethanol infusion — Vein of Marshall ethanol infusion performed during the radiofrequency catheter ablation of persistent or long-standing persistent atrial fibrillation.

SUMMARY:
The study is a prospective, randomized, single-blind clinical trial aiming to compare two method in guidance of Vein of Marshall ethanol infusion (VOMEI), i.e., the conventional fluoroscopy-guided VOMEI and UNIVU-guided VOMEI.

DETAILED DESCRIPTION:
A total of 100 participants with persistent or longstanding persistent AF who undergo radiofrequency catheter ablation will be randomized assigned to two groups at 1:1 ratio to receive Vein of Marshall ethanol infusion (VOMEI).

Group 1: VOMEI guided by fluroscopy alone Group 2: VOMEI guided by fluoroscopy and CARTO UNIVU The intraprocedural major endpoints are the change in low-voltage area led by VOMEI (efficacy endpoint) and procedural complications (safety endpoint). The longterm major endpoint is the recurrence of atrial tachyarrhythmia between 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Sympathetic atrial fibrillation without previous ablation
* Persistent or long-standing persistent AF
* Patients' willing to undergo catheter ablation and VOMEI

Exclusion Criteria:

* Left atrial or left atrial appendage thrombus
* LVEF <30%
* Cardiac surgery within 90 days
* Myocardial infarction within 90 days
* PCI or PTCA within 90 days
* Thromboembolic events within 90 days, including stroke, pulmonary embolism, systemic embolism
* Atrial myxoma
* Congenital heart disease
* Pregnant or pregnant plan
* Acute or severe infection
* Creatine> 221 μmol/L, or GFR <30 ml/min/1.73 m.
* Unstable angina
* Blood-clotting or bleeding disorder
* Contraindication to anticoagulation
* Life expectancy less than 1 year
* Uncontrolled heart failure
* Uncontrolled malignant tumor
* Malformation of femoral vascular access
* Without consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of low-voltage or scar area before and after VOMEI | During the procedure
  Left atrial voltage mapping will be performed before and after VOMEI. The low-voltage area or scar area will be mesured and compared before and after VOMEI
Procedural complications | within 72 hours
  Including cardiac tamponade, stroke, systemic embolism, major bleeding, acute coronary syndrome, acute heart failure, and death.
Recurrence of atrial tachyarrhythmias | 3 to 12 months
  Including recurrence of atrial fibrillation, atrial flutter, and atrial tachycardia

SECONDARY OUTCOMES:
Rates of mitral isthmus block | During the procedure
  bidirectional block of mitral isthmus
New low-voltage or scar area outside mitral isthmus and left pulmonary ridge | During the procedure
  New low-voltage or scar area after VOMEI outside the targeted regions
Rates of VOMEI incomplete | During the procedure
  Any reason leading to incomplete VOMEI
X ray exposure time | During the procedure
  Procedure-related temporal parameters
procedure time | During the procedure
  Procedure-related temporal parameters
radiofrequency ablation time | During the procedure
  Procedure-related temporal parameters
Rates of intraprocedural termination of atrial fibrillation (not achieved by cardioversion) | During the procedure
  Termination of atrial fibrillation without cardioversion
Burden of atrial tachyarrhythmia | 12 months
  Evaluation by Holder monitoring at 12 months
Recurrence of atrial flutter | 3 to 12 months
  recurrence of atrial flutter > 30 second by ECG or Holder monitoring
Volume of ethanol and contrast agent used | During the procedure
  ethanol volume, contrast agent volume used during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jian Sun, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China